CLINICAL TRIAL: NCT00253942
Title: A Randomized, Double-Blind, Histamine-Controlled, Phase 3 Study to Determine the Safety and Efficacy of Bee Venom in the Treatment of Knee Osteoarthritis
Brief Title: Safety and Efficacy Study of Bee Venom to Treat Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rheumatology Therapeutics Medical Center (Other)
Collaborators: Kochan Institute for Healing Arts Research (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OABVTKNEE-001
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-10

CONDITIONS: Persons With Mild to Moderate Knee Osteoarthritis

INTERVENTIONS:
Procedure: Injecting bee venom as a treatment for OA

SUMMARY:
Study wishes to determine if the use of injectable bee venom is a safe and effective treatment for persons with mild to moderate knee Osteoarthritis and would result in decreased report of pain and discomfort, increased function during daily activities, decrease use of analgesic meds, and improvement in walking and climbing steps. We will be using histamine as a control. 40 subjects will be enrolled in a 3:1 allocation ratio between bee venom and histamine. Each injection of bee venom dosage will consist of 100 micrograms of dried bee venom in 0.1 ml. of 0.5% preservative free Xylocaine. The histamine dosage will consist of .0025 milligrams of histamine in 0.5% preservative free Xylocaine. Subjects will visit the study center for 14 visits over an 18 week span. The clinical hypothesis is that bee venom is an effective treatment for Osteoarthritis and will reduce pain and discomfort, increase range of motion, increase daily function, decrease walking and stair climbing time, and decrease the need of analgesic medication for a period of time beyond treatment (after the study has concluded.) The clinical safety hypothesis is that for persons not allergic to bee venom (patients allergic will not be allowed to enter into the study) the side effects will be small. The most common side effects for bee venom and histamine will be redness and itchiness which will be tolerable and safe.

ELIGIBILITY:
Inclusion Criteria:

* Meet clinical criteria for Osteoarthritis in one knee
* Morning stiffness less than 30 minutes duration
* VAS pain level of 4 to 8 on a 0 to 10 scale when walking
* Older than 35 years of age
* On a stable dose of medication or none at all due to intolerance
* Ability to tolerate Acetaminophen as their only pain medication for the entire study
* Ability to read, understand, and give informed consent and sign the informed consent form

Exclusion Criteria:

* Allergy to bee venom or histamine
* Allergy to Lidocaine
* Any type of inflammatory arthritis such as RA, SLE, Psoriatic
* Fibromyalgia or any pain problem that requires the use of pain medication or anti-inflammatory
* Depression or any condition that interferes with memory or critical analysis
* History of prolotherapy, bee venom therapy, or injection of hyaluronic acid or cortisone within the last 3 months
* Osteoarthritis of the hip, ankle, or any condition that interferes with walking 50 ft. or up and down stairs
* Elevated CRP, SED rate
* Recent injury to the knee which is causing pain or functional problems
* Any previous invasive procedure on the study knee
* Inability to understand the informed consent form or refusal to sign it
* Cardiac disease interfering with ability to get epinephrine
* VAS pain level greater than 8 on a 0 to 10 scale when walking
* Inability to stop anti-inflammatory medication for the entire study and use only Acetaminophen
* Taking beta blockers
* Taking chronic anti-histamines

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-11

PRIMARY OUTCOMES:
Change in Visual Analog Scale
Change in Knee Injury and Osteoarthritis Outcome Score
Change in use of analgesic meds after 6 weeks of treatment
Change in 50 ft. walk and 4 step up/down climb time

SECONDARY OUTCOMES:
Adverse event incidence
Baseline and visit 12 laboratory assessments
Change in tenderness and motion

CONTACTS AND LOCATIONS:
Overall Officials: Boris Ratiner, MD, Principal Investigator — Medical Director of Rheumatology Therapeutics Medical Center; Andrew Kochan, MD, Principal Investigator — Medical Director of Kochan Institute for Healing Arts Research
Locations (2):
- United States (2):
  - Kochan Institute for Healing Arts Research, Encino, California
  - Rheumatology Therapeutics Medical Center, Tarzana, California